CLINICAL TRIAL: NCT01472471
Title: Urinary 8-isoprostane is Elevated in Acute Childhood Asthma
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Other Study IDs: 171086-4
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Childhood Asthma; Oxidative Stress
Keywords: Childhood Asthma; Oxidative stress; Urinary 8-isoprostane

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- acute asthmatic children: Children hospitalized with a diagnosis of acute asthma exacerbation
- stable asthmatic children: Children with a history of asthma currently asymptomatic

SUMMARY:
Oxidative stress is seen in children with asthma, but is hard to measure. The investigators exploring the utility of using a commercially available assay to measure oxidative stress in the urine in asthmatics. Additionally, the investigators will attempt to prove that oxidative stress is higher in children with acute asthma compared to those with stable asthma and that this stress is also higher in children with more severe clinical asthma exacerbations compared to less severe ones.

ELIGIBILITY:
Inclusion Criteria:

Group 1

1. Patients aged 4-18 years
2. Known stable asthmatics on no medications or with no medication changes in 3 weeks prior to enrollment
3. No asthma hospitalizations in past 3 months
4. Parent available to consent

Group 2

1. Patients aged 4-18
2. Known asthmatic, admitted to Stony Brook University Hospital for status asthmaticus
3. Parent available to consent

Exclusion Criteria:

1. Any child with documented fever within 24 hours of study entry
2. Any child with a known current history of tracheo- or bronchomalacia
3. Any child with known clinical or laboratory evidence of shock (see below)
4. Any child with history of documented immunodeficiency, rheumatologic disease, cystic fibrosis, or renal dysfunction (see below)
5. Any child with a current or recent (less than 1 year) history of tracheostomy
6. Any child with a known genetic abnormality
7. Any pregnant child
8. Any child with a history of autism
9. Any child whose parent/caregiver is unable to give informed consent

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Group 1:
  25 subjects will be recruited from among the children seen at the Stony Brook University Pediatric Pulmonary and Allergy Clinic.
  Group 2 25 subjects will be recruited from among the children admitted to Stony Brook University Hospital with a diagnosis of acute asthma exacerbation or reactive airway disease from Monday at 12 AM to Friday at 5 PM.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
We expect to see increased urinary 8-isoprostane in acute pediatric asthmatics | Urinary 8-isoprostane levels were measured at the end of subject recruitment

SECONDARY OUTCOMES:
We expect urinary 8-isoprostane levels to be higher with increased pediatric asthma severity. | This was calculated at the end of patient recruitment, after urinary 8-isoprostane levels were obtained

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Sloniewsky, MD, Principal Investigator — Long Island Children's Hospital at Stony Brook
Locations (1):
- Long Island Children's Hospital at Stony Brook, Stony Brook, New York, United States